CLINICAL TRIAL: NCT02918019
Title: A Phase IIb, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Dose-Ranging Study to Assess the Efficacy and Safety of MSTT1041A in Patients With Uncontrolled Severe Asthma
Brief Title: A Study to Assess the Efficacy and Safety of MSTT1041A in Participants With Uncontrolled Severe Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GB39242; 2016-001549-13 (EudraCT Number)
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Results first posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — astegolimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MSTT1041A 210 mg (Experimental): Participants will receive MSTT1041A 210 milligrams (mg), subcutaneously every 4 weeks from randomization through Week 50.
  Interventions: Drug: MSTT1041A
- MSTT1041A 490 mg (Experimental): Participants will receive MSTT1041A 490 mg, subcutaneously every 4 weeks from randomization through Week 50.
  Interventions: Drug: MSTT1041A
- MSTT1041A 70 mg (Experimental): Participants will receive MSTT1041A 70 mg, subcutaneously every 4 weeks from randomization through Week 50.
  Interventions: Drug: MSTT1041A
- Placebo (Placebo Comparator): Participants will receive placebo matched with MSTT1041A, subcutaneously every 4 weeks from randomization through Week 50.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MSTT1041A — MSTT1041A will be administered as subcutaneous injections.
  Other Names: RO7187807
  Arms: MSTT1041A 210 mg; MSTT1041A 490 mg; MSTT1041A 70 mg
Drug: Placebo — Placebo matched with MSTT1041A.
  Arms: Placebo

SUMMARY:
This is a Phase IIb, randomized, placebo-controlled, double-blind, multicenter, multi-arm study which will evaluate efficacy, safety, and pharmacokinetic of MSTT1041A compared with placebo as add-on therapy in participants with severe, uncontrolled asthma who are receiving medium- or high-dose inhaled corticosteroid (ICS) therapy and at least one of the following additional controller medications: long-acting beta-agonists (LABA), leukotriene modifier (LTM), long-acting muscarinic antagonist (LAMA), or long-acting theophylline preparation. The total duration of this study for each participant is approximately 70 weeks including screening, run-in, treatment, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 18 to 38 kilogram/square meter (kg/m^2) and weight >= 40 kg at screening
* Documented physician-diagnosed asthma
* On high dose inhaled corticosteroid (ICS) therapy plus at least one additional allowed controller medication
* Forced expiratory volume in 1 second (FEV1) of 40% to 80% of predicted
* Evidence of uncontrolled asthma
* Use of contraceptive measures

Exclusion Criteria:

* Diagnosis of mimics of asthma
* Diagnosis of occupational asthma, aspirin-sensitive asthma, asthma chronic obstructive pulmonary disease overlap syndrome, or bronchiolitis, as determined by the investigator
* Pregnant or lactating, or intending to become pregnant during the study or within 20 weeks after the last dose of MSTT1041A
* Recent history of smoking
* History or evidence of substance abuse that would pose a risk to participants safety, interfere with the conduct of the study, have an impact on the study results
* Asthma exacerbation within 4 weeks prior to screening
* Intubation for respiratory failure due to asthma within 12 months prior to screening
* Comorbid conditions that may interfere with evaluation of investigational medicinal product
* Known sensitivity to any of the active substances or their excipients to be administered during dosing
* Positive pregnancy test

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (138):
- United States (43):
  - Alabama Allergy & Asthma, Birmingham, Alabama
  - Del Sol Research Management, Tucson, Arizona
  - Kern Allergy Med Clinic, Inc., Bakersfield, California
  - Allergy & Asthma Care Center of Southern California, Long Beach, California
  - CA Allergy & Asthma Med Grp; Medical Group, Inc., Los Angeles, California
  - Jonathan Corren MD, Inc., Los Angeles, California
  - Office of Robert N Wolfe MD, Los Angeles, California
  - Advances in Medicine, Rancho Mirage, California
  - Allergy & Asthma Consultants, Redwood City, California
  - Bensch Research Associates, Stockton, California
  - Allergy and Asthma Clinical Research, Inc., Walnut Creek, California
  - IMMUNOe Research Centers, Centennial, Colorado
  - Asthma & Allergy; Associates, P.C., Colorado Springs, Colorado
  - Western States Clinical Research, Inc, Wheat Ridge, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - Emerald Coast Research Associates, Panama City, Florida
  - Florida Premier Research Institute, Winter Park, Florida
  - Atlanta Allergy & Asth Clin PC, Stockbridge, Georgia
  - Asthma & Allergy of Idaho, Twin Falls, Idaho
  - Asthma, Allergy & Sinus Center, Baltimore, Maryland
  - Chesapeake Clinical Research Inc - CRN, Baltimore, Maryland
  - Genesis Clinical Research & Consulting, LLC, Fall River, Massachusetts
  - Infinity Medical Research Inc, North Dartmouth, Massachusetts
  - Midwest Clinical Research LLC, St Louis, Missouri
  - The Allergy and Asthma Center, Bellevue, Nebraska
  - Montefiore Medical Center, The Bronx, New York
  - American Health Research Inc., Charlotte, North Carolina
  - Allergy & Respiratory Center, Canton, Ohio
  - Integrity People Services Research Company, Oklahoma City, Oklahoma
  - Vital Prospects Clin Res Pc, Tulsa, Oklahoma
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Asthma & Allergy Physicians of Rhode Island Clinical Research Institute (AAPRI CRI), Warwick, Rhode Island
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Clinical Research Solutions PC, Knoxville, Tennessee
  - Meharry Medical College; Clinical Trials Office, Nashville, Tennessee
  - TTS Research, Boerne, Texas
  - Elliot J. Ginchansky, MD, PA, Dallas, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Metroplex Pulmonology & Sleep Center, McKinney, Texas
  - Allergy & Asthma Research Center, San Antonio, Texas
  - Allergy Associates of Utah, Murray, Utah
  - Commonwealth Clinical Research Specialists, Richmond, Virginia
  - Washington Univ School of Med, Seattle, Washington
- Argentina (10):
  - Fundacion Cidea, Buenos Aires
  - INAER, Buenos Aires
  - Fundacion Scherbovsky, Mendoza
  - INSARES, Mendoza, Mendoza City
  - Centro Respiratorio Quilmes, Quilmes
  - Instituto Especialidades de la Salud Rosario, Rosario
  - Instituto de Diagnóstico ABC; Servicio de Investigación de Patologías Alérgicas, Rosario
  - Centro Modelo de Cardiologia, San Miguel de Tucumán
  - Investigaciones en Patologias Respiratorias, San Miguel de Tucumán
  - CEMER Centro Medico de Enfermedades Respiratorias, Vicente López
- Belgium (2):
  - Cliniques Universitaires St-Luc, Brussels
  - Private Practice Dr Jean Benoit Martinot, Erpent
- Bulgaria (12):
  - Military Medical Academy HBAT, Pleven
  - SHATPPD Dr. Dimitar Gramatikov, Ruse Ltd., Rousse
  - Medical Centre Mladost Med 1 EOOD, Sofia
  - First MHAT; Clinic of Neurology, Sofia
  - Fifth MHAT - Sofia EAD, Sofia
  - National Multiprofile Hospital Tsar Boris III, Sofia
  - Specialised Hospital for Active Treatment of Pulmonary Deseases "Sv. Sofia", Third Clinic for Non-Sp, Sofia
  - Uni. Multiprofile Hosp. for Active Treatment-Aleksandrovska, Sofia
  - Medical Center N.I. Pirogov EOOD, Sofia
  - Alitera - Med - Medical Center EOOD, Sofia
  - Medical Center "Nov Rehabilitatsionen Tsentar", EOOD, Stara Zagora
  - Medical Center Tara OOD, Veliko Tarnovo
- Canada (5):
  - Aggarwal and Associates, Brampton, Ontario
  - Cheema Research, Mississauga, Ontario
  - Inspiration Research, Toronto, Ontario
  - Anil Dhar Professional Medicine Corporation, Windsor, Ontario
  - C.I.C. Mauricie, Trois-Rivières, Quebec
- Czechia (5):
  - MediTrial s.r.o., Jindřichův Hradec
  - EUC Klinika Ostrava a.s., Ostrava-Poruba
  - Ordinace pro tuberkulozu a respiracni nemoci, Strakonice
  - KASMED s.r.o., Tábor
  - Alergologie Teplice, s.r.o., Teplice
- Germany (4):
  - Pneumologisches Forschungsinstitut Hohegeest, Geesthacht
  - POIS Leipzig Gbr, Leipzig
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Medizinische Klinik, Pneumologie, Mainz
  - Universitatsklinikum Munster, Münster
- New Zealand (2):
  - Greenlane Clinical Centre, Auckland
  - Medical Research Institute of New Zealand, Wellington
- Peru (6):
  - Clinica Internacional, Lima
  - Abk Reuma Srl- Medicentro, Lima
  - Clinica Ricardo Palma; THORAX, Lima
  - Instituto Peruano de Investigacion en Ciencias Medicas, Lima
  - Clinica San Borja, Lima
  - Hospital Santa Rosa Piura, Piura
- Poland (10):
  - Centrum Medycyny Oddechowej Robert M. Mróz, Bialystok
  - Centrum Medyczne ALL-MED, Krakow
  - Malopolskie Centrum Alergologii, Krakow
  - Niepubliczny Zaklad Opieki Zdrowotnej Centrum Medyczne ProMiMed sp z o.o. sp.k., Krakow
  - SPZOZ Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz
  - Specjalistyczna Poradnia Pulmonologiczna, Ostrów Wielkopolski
  - Przedsiebiorstwo Podmiotu Leczniczego Poradnie Specjalistyczne MAGMED, Radom
  - ALERGO-MED Specjalistyczna Przychodnia Lekarska Sp. z o. o, Tarnów
  - Ewa Pisarczyk-Bogacka Specjalistyczna Praktyka Lekarska, Wroclaw
  - NZOZ Lekarze Specjaliści J. Małolepszy i Partnerzy, Wroclaw
- Romania (5):
  - Theramed SRL, Brasov
  - Spitalul Clinic de Pneumoftiziologie Leon Daniello Cluj-Napoca, Sectia Clinica Pneumologie I, Cluj-Napoca
  - Spitalul Clinic de Boli Infectioase si Pneumoftiziologie Victor Babes Craiova, Craiova
  - Fundatia CardioPrevent, Timișoara
  - Dr. Victor Babes Pneumology and Infectious Diseases Clinical Hospital, Timișoara
- Russia (13):
  - Clinical Emergency Hospital n.a.N.V. Soloviev, Yaroslavl, Moscow Oblast
  - LLC - ABC Medicina, Moscow, Sankt-Peterburg
  - City Hospital #5, Barnaul
  - Municipal Healthcare Institution City Clinical Hospital #3 named after M.A. Podgorbunskogo, Kemerovo
  - I.M. Sechenov Moscow State Medical University the Ministry of Health and Social Development of RF, Moscow
  - Novosibirsk Municipal Clinical Hospital For Emergency Medicine #2, Novosibirsk
  - City Clinical Hospital #2, Novosibirsk
  - Ryazan State Medical University Named after I.P.Pavlov, Ryazan
  - Clinic Reavita LLC, Saint Petersburg
  - SHI Ctr Occupational Pathology, Saint Petersburg
  - St. Petersburg State Medical University n.a. I.P. Pavlov, Saint Petersburg
  - City Hospital #40 of Resort Administrative District, Saint Petersburg
  - Siberian State Medical University, Tomsk
- South Africa (5):
  - Tiervalei Trial Centre, Cape Town
  - University of Cape Town Lung Institute; Lung Clinical Research, Cape Town
  - St Augustines Hospital; Infectoilogy, Durban
  - Vawda Z.Fa Practice, Durban
  - Aliwal Shoal Medical Center, eMkhomazi
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Ukraine (13):
  - Regional Municipal Institution Chernivtsi Regional Clinical Hospital, Chernivtsi, Chernihiv Governorate
  - Municipal institution; City hospital #1; Department of Therapy, Zaporizhzhia, Kherson Governorate
  - Kyiv City Tuberculosis Hospital #1; Department of Differential Diagnosis of Lung Diseases, Kyiv, KIEV Governorate
  - Public Institution City Clinical Hospital # 6 of Dnipropetrovsk Regional Board, Dnipro
  - Ukrainian State Institute of Medical and Social Problems of Disability, Dnipropetrovsk
  - Regional Phthisiology and Pulmonology Center, Ivano-Frankivsk
  - SI Institute of Therapy n.a. L.T. Mala of National Academy of Medical Sciences of Ukraine, Kharkiv
  - SI National Institute of Phthisiology and Pulmonology n.a. F.G.Yanovskyi under NAMS of Ukraine, Kyiv
  - Municipal Institution of Kyiv Regional Council Kyiv Regional Clinical Hospital, Kyiv
  - Kyiv City Clinical Hospital #8, Kyiv
  - City Hospital #1, Mykolaiv
  - Municipal Institution Odesa Regional Clinical Hospital, Odesa
  - Small Business Private Enterprise Medical Centre Pulse, Vinnytsia

REFERENCES:
- [Derived] Yin Z, Zhou Y, Turnquist HR, Liu Q. Neuro-epithelial-ILC2 crosstalk in barrier tissues. Trends Immunol. 2022 Nov;43(11):901-916. doi: 10.1016/j.it.2022.09.006. Epub 2022 Oct 14. PMID 36253275
- [Derived] Kelsen SG, Agache IO, Soong W, Israel E, Chupp GL, Cheung DS, Theess W, Yang X, Staton TL, Choy DF, Fong A, Dash A, Dolton M, Pappu R, Brightling CE. Astegolimab (anti-ST2) efficacy and safety in adults with severe asthma: A randomized clinical trial. J Allergy Clin Immunol. 2021 Sep;148(3):790-798. doi: 10.1016/j.jaci.2021.03.044. Epub 2021 Apr 16. PMID 33872652

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants with severe, uncontrolled asthma receiving medium- or high-dose inhaled corticosteroid (ICS) therapy and at least one additional controller medication.
Pre-assignment Details: Fifteen participants were randomized in error and only 502 of 517 participants received at least one dose of study drug. The 15 participants were not included in further analysis.
Groups:
- Placebo: Participants received subcutaneous (SC) placebo matched to astegolimab (MSTT1041A) at randomization (Week 2), Week 6, and every 4 weeks (Q4W) thereafter through Week 50.
- Astegolimab (MSTT1041A) 70mg: Participants received 70mg of SC astegolimab (MSTT1041A) at randomization (Week 2), Week 6, and every 4 weeks (Q4W) thereafter through Week 50.
- Astegolimab (MSTT1041A) 210mg: Participants received 210mg of SC astegolimab (MSTT1041A) at randomization (Week 2), Week 6, and every 4 weeks (Q4W) thereafter through Week 50.
- Astegolimab (MSTT1041A) 490mg: Participants received 490mg of SC astegolimab (MSTT1041A) at randomization (Week 2), Week 6, and every 4 weeks (Q4W) thereafter through Week 50.
Period: Overall Study
Arm/Group | Placebo | Astegolimab (MSTT1041A) 70mg | Astegolimab (MSTT1041A) 210mg | Astegolimab (MSTT1041A) 490mg
Started | 127 | 127 | 126 | 122
Completed | 121 | 117 | 117 | 113
Not Completed | 6 | 10 | 9 | 9
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1
Not completed — Principal investigator request | 0 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 3 | 2 | 0
Not completed — Protocol deviation | 1 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 3 | 4 | 6 | 4
Not completed — Adverse Event | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Astegolimab (MSTT1041A) 70mg | Astegolimab (MSTT1041A) 210mg | Astegolimab (MSTT1041A) 490mg | Total
Number analyzed (Participants) | 127 | 127 | 126 | 122 | 502
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (12.2) | 52.4 (11.9) | 52.5 (12.0) | 51.4 (12.0) | 51.9 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 81 | 90 | 79 | 332
  Male | 45 | 46 | 36 | 43 | 170
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 19 | 15 | 14 | 66
  Not Hispanic or Latino | 109 | 108 | 110 | 108 | 435
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 5 | 8 | 4 | 22
  Asian | 6 | 4 | 4 | 9 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 9 | 6 | 6 | 29
  White | 107 | 105 | 108 | 102 | 422
  More than one race | 1 | 4 | 0 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Absolute Change in Pre-Bronchodilator Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 measures how much air a person can exhale during the first second of a forced breath.
  Adjusted means are reported.
Time Frame: Baseline to Week 54
Measure: Mean (95% Confidence Interval); unit: Milliliters (mL)
Arm/Group | Placebo | Astegolimab (MSTT1041A) 70mg | Astegolimab (MSTT1041A) 210mg | Astegolimab (MSTT1041A) 490mg
Number analyzed (Participants) | 120 | 117 | 115 | 113
Milliliters (mL) | 107 (47) [47 to 167] | 130 (70) [70 to 191] | 154 (93) [93 to 215] | 172 (110) [110 to 234]

2. Secondary Outcome: Time to First Asthma Exacerbation
Description: Asthma exacerbation was defined as new or increased asthma symptoms (wheezing, coughing, dyspnea, chest tightness, and/or nighttime awakenings due to these symptoms) that result in one or both of the following: Hospitalization or emergency department visit with administration of systemic corticosteroid treatment; Treatment with systemic corticosteroids for at least 3 days, or a long-acting depot corticosteroid preparation with a therapeutic effectiveness of at least 3 days.
Time Frame: 52 Weeks
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo | Astegolimab (MSTT1041A) 70mg | Astegolimab (MSTT1041A) 210mg | Astegolimab (MSTT1041A) 490mg
Number analyzed (Participants) | 127 | 127 | 126 | 122
Weeks | NA [46.6 to NA] — Value not estimable due to insufficient no. of participants with event | NA [NA to NA] — Value not estimable due to insufficient no. of participants with event | NA [NA to NA] — Value not estimable due to insufficient no. of participants with event | NA [NA to NA] — Value not estimable due to insufficient no. of participants with event

3. Secondary Outcome: Achievement in Improvement in Standardized Asthma Quality-of-Life Questionnaire (AQLQ(S)) Score
Description: The AQLQ measures the functional problems (physical, emotional, social, and occupational) most troublesome to adults (17-70 years) with asthma. There are 32 questions in 4 domains - symptoms, activity limitation, emotional function, and environmental stimuli - scored on a 7 point scale, with 7= no impairment and 1= severely impaired. For this study, improvement achievement was defined as an increase of at least 0.5 points from baseline to week 54.
  Adjusted rates are reported.
Time Frame: Week 54
Measure: Number; unit: Percentage
Arm/Group | Placebo | Astegolimab (MSTT1041A) 70mg | Astegolimab (MSTT1041A) 210mg | Astegolimab (MSTT1041A) 490mg
Number analyzed (Participants) | 116 | 116 | 115 | 112
Percentage
  Week 54 - Responder | 55.3 | 64.8 | 61.3 | 68.9
  Week 54 - Non-responder | 44.7 | 35.2 | 38.7 | 31.1

4. Secondary Outcome: Absolute Change in Patient-Reported Use of Short-Acting Rescue Therapy
Description: Adjusted mean values are all equal to zero.
Time Frame: Baseline to Week 54
Measure: Mean (95% Confidence Interval); unit: Usage
Arm/Group | Placebo | Astegolimab (MSTT1041A) 70mg | Astegolimab (MSTT1041A) 210mg | Astegolimab (MSTT1041A) 490mg
Number analyzed (Participants) | 107 | 106 | 102 | 99
Usage | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

5. Secondary Outcome: Proportion of Weeks Without Patient-Reported Asthma-Related Nighttime Awakenings
Description: The adjusted mean proportion of weeks without a nighttime awakening from baseline through week 54 are reported. The proportion of weeks is expressed as a percentage.
Time Frame: Baseline through Week 54
Measure: Mean (95% Confidence Interval); unit: Percentage of weeks
Arm/Group | Placebo | Astegolimab (MSTT1041A) 70mg | Astegolimab (MSTT1041A) 210mg | Astegolimab (MSTT1041A) 490mg
Number analyzed (Participants) | 127 | 126 | 126 | 122
Percentage of weeks | 0.4 [-0.7 to 1.5] | 0.4 [-0.7 to 1.5] | 0.3 [-0.7 to 1.3] | 0.3 [-0.7 to 1.3]

6. Secondary Outcome: Absolute Change in Patient-Reported Daytime Asthma Symptom Severity as Measured by the Asthma Daily Symptom Diary (ADSD)
Description: The ADSD is a 6-item daily measure of asthma symptom severity that assesses three core categories of asthma symptoms: breathing symptoms, chest symptoms, and cough. Symptoms are rated at their worst using an 11-point numeric rating scale ranging from 0 (no symptoms) to 10 (the worst symptoms imaginable).
  Adjusted means are reported.
Time Frame: Baseline to Week 54
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | Astegolimab (MSTT1041A) 70mg | Astegolimab (MSTT1041A) 210mg | Astegolimab (MSTT1041A) 490mg
Number analyzed (Participants) | 126 | 124 | 125 | 122
Scores on a scale | -1 [-2 to -1] | -2 [-2 to -1] | -1 [-2 to -1] | -1 [-2 to -1]

7. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline to Week 54
Measure: Number; unit: Percentage
Arm/Group | Placebo | Astegolimab (MSTT1041A) 70mg | Astegolimab (MSTT1041A) 210mg | Astegolimab (MSTT1041A) 490mg
Number analyzed (Participants) | 127 | 127 | 126 | 122
Percentage | 77.2 | 70.9 | 72.2 | 72.1

8. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADAs)
Description: The prevalence of ADAs at baseline was defined as the proportion of the evaluable participant population in a study that is ADA positive at baseline.
Time Frame: Baseline
Measure: Number; unit: Percentage
Arm/Group | Placebo | Astegolimab (MSTT1041A) 70mg | Astegolimab (MSTT1041A) 210mg | Astegolimab (MSTT1041A) 490mg
Number analyzed (Participants) | 124 | 126 | 126 | 121
Percentage | 5.6 | 0.8 | 1.6 | 1.7

9. Secondary Outcome: Serum Concentration of Astegolimab (MSTT1041A)
Time Frame: Weeks 26 and 54
Population: The analysis population consisted of all PK-evaluable participants with at least one serum PK collected for the given treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Astegolimab (MSTT1041A) 70mg | Astegolimab (MSTT1041A) 210mg | Astegolimab (MSTT1041A) 490mg
Number analyzed (Participants) | 125 | 126 | 117
ug/mL
  Week 26 pre-dose: number analyzed (Participants) | 120 | 113 | 113
  Week 26 pre-dose | 4.75 (123.3) | 16.9 (167.3) | 40.5 (161.2)
  Week 54: number analyzed (Participants) | 116 | 117 | 111
  Week 54 | 4.47 (144.1) | 17.4 (155.4) | 38.7 (226.4)

10. Secondary Outcome: Percentage of Participants With Treatment-Emergent ADAs
Description: The incidence of ADAs at post-baseline timepoints was defined as the proportion of the study population found to have developed treatment-emergent ADAs.
Time Frame: From baseline to the first appearance of ADAs at any point post-baseline (up to Week 54)
Measure: Number; unit: Percentage
Arm/Group | Placebo | Astegolimab (MSTT1041A) 70mg | Astegolimab (MSTT1041A) 210mg | Astegolimab (MSTT1041A) 490mg
Number analyzed (Participants) | 126 | 125 | 123 | 120
Percentage | 7.1 | 9.6 | 8.9 | 3.3

11. Primary Outcome: Reduction in Rate of Asthma Exacerbations
Description: Asthma exacerbation was defined as new or increased asthma symptoms (wheezing, coughing, dyspnea, chest tightness, and/or nighttime awakenings due to these symptoms) that result in one or both of the following: Hospitalization or emergency department visit with administration of systemic corticosteroid treatment; Treatment with systemic corticosteroids for at least 3 days, or a long-acting depot corticosteroid preparation with a therapeutic effectiveness of at least 3 days.
  Adjusted rates for the overall mITT population (all participants that received at least one dose of study drug) were estimated using Poisson regression and adjusted for blood eosinophil level at the first visit, the number of asthma exacerbations requiring systemic corticosteroids in the 12 months prior to study entry, the total daily ICS dose at the first visit, and geographic region, with patient time at risk used as an offset term.
Time Frame: Baseline to Week 54
Measure: Number; unit: Number of asthma exacerbations per year
Arm/Group | Placebo | Astegolimab (MSTT1041A) 70mg | Astegolimab (MSTT1041A) 210mg | Astegolimab (MSTT1041A) 490mg
Number analyzed (Participants) | 120 | 127 | 126 | 122
Number of asthma exacerbations per year | 0.74 | 0.47 | 0.58 | 0.42
Statistical Analysis 1: Comparison: Astegolimab (MSTT1041A) 490mg; Test type: Other; p = 0.0049, Poisson regression; Rate Ratio = 0.57, 95% CI 2-sided [0.39 to 0.84]
Statistical Analysis 2: Comparison: Astegolimab (MSTT1041A) 210mg; Test type: Other; p = 0.1838, Poisson regression; Rate Ratio = 0.78, 95% CI 2-sided [0.54 to 1.12]
Statistical Analysis 3: Comparison: Astegolimab (MSTT1041A) 70mg; Test type: Other; p = 0.0144, Poisson regression; Rate Ratio = 0.63, 95% CI 2-sided [0.44 to 0.91]

ADVERSE EVENTS:
Time Frame: Baseline to Week 54
Arm/Group | Placebo | Astegolimab (MSTT1041A) 70mg | Astegolimab (MSTT1041A) 210mg | Astegolimab (MSTT1041A) 490mg
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/127 | 1/126 | 1/122
Serious Adverse Events (participants affected / at risk) | 8/127 | 14/127 | 9/126 | 6/122
Other Adverse Events (participants affected / at risk) | 76/127 | 65/127 | 75/126 | 68/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=127) | Astegolimab (MSTT1041A) 70mg (N=127) | Astegolimab (MSTT1041A) 210mg (N=126) | Astegolimab (MSTT1041A) 490mg (N=122)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 4 (4) | 1 (1)
Chronic rhinosinusitis with nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=127) | Astegolimab (MSTT1041A) 70mg (N=127) | Astegolimab (MSTT1041A) 210mg (N=126) | Astegolimab (MSTT1041A) 490mg (N=122)
Injection site reaction (General disorders) | 1 (3) | 10 (38) | 8 (23) | 6 (107)
Influenza (Infections and infestations) | 5 (5) | 2 (2) | 2 (2) | 7 (7)
Nasopharyngitis (Infections and infestations) | 13 (18) | 12 (21) | 21 (30) | 16 (23)
Rhinitis (Infections and infestations) | 7 (8) | 7 (11) | 3 (3) | 2 (3)
Sinusitis (Infections and infestations) | 3 (3) | 7 (9) | 3 (3) | 5 (7)
Upper respiratory tract infection (Infections and infestations) | 12 (19) | 9 (10) | 8 (9) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 7 (7) | 4 (5) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 5 (5) | 5 (5) | 4 (4)
Headache (Nervous system disorders) | 6 (6) | 8 (10) | 6 (7) | 14 (20)
Asthma (Respiratory, thoracic and mediastinal disorders) | 58 (108) | 42 (68) | 53 (83) | 39 (61)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/19/NCT02918019/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT02918019/SAP_001.pdf